CLINICAL TRIAL: NCT00004179
Title: Chimeric Anti-CD20 Monoclonal Antibody (Mabthera) in Remission Induction and Maintenance Treatment of Relapsed Follicular Non-Hodgkin's Lymphoma: A Phase III Randomized Clinical Trial - Intergroup Collaborative Study
Brief Title: Combination Chemotherapy With or Without Rituximab in Treating Patients With Relapsed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Lymphoma Trials Office (Other); Stichting Hemato-Oncologie voor Volwassenen Nederland (Other); Australasian Leukaemia and Lymphoma Group (Other); NCIC Clinical Trials Group (Network); Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-20981; EORTC-20981 (Other: EORTC); ALLG-NHLLOW4 (Other: ALLG); BNLI-EORTC-20981 (Other: BNLI); HOVON-H039 (Other: HOVON); CAN-NCIC-LY7 (Other: NCIC CTG); NORDIC-EORTC-20981 (Other: NLG)
Record Dates: First submitted 2000-01-21; First posted 2003-01-27 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; VAP-cyclo protocol; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

INTERVENTIONS:
Biological: rituximab
Drug: CHOP regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known whether chemotherapy is more effective with or without rituximab for relapsed non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying combination chemotherapy and rituximab to see how well they work compared to combination chemotherapy alone in treating patients with relapsed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate and quality of remission in patients with relapsed follicular non-Hodgkin's lymphoma treated with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) with or without rituximab.
* Compare the event-free survival and overall survival of patients treated with these regimens.
* Determine the effect of rituximab as maintenance therapy on progression-free survival of these patients.

OUTLINE: This is a randomized, multicenter study.

* Induction: Patients are randomized to one of two treatment arms. Patients are stratified according to participating center, prior treatment with purine analogues, age, number of prior induction treatments and best response obtained (complete vs partial remission vs no change/progressive disease), time since diagnosis (less than 2 years vs more than 2 years), and bulky disease (less than 10 cm vs greater than 10 cm).

  * Arm I (closed as of 12/20/04): Patients receive induction chemotherapy comprising cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5 (CHOP chemotherapy). Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive CHOP chemotherapy as in arm I. Rituximab IV is administered 1 hour after prednisone and before the IV drugs.
* Maintenance: Patients who achieve partial or complete remission are then randomized to one of two treatment arms. Patients are stratified according to rituximab administration during induction (yes vs no), quality of the response (complete vs partial remission vs no change/progressive disease), and participating center.

  * Arm I: Patients receive no further therapy.
  * Arm II: Beginning 8 weeks after the last CHOP course, patients receive rituximab IV once every 3 months for up to 2 years in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 4 months thereafter.

PROJECTED ACCRUAL: A total of 752 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven stage III or IV follicular non-Hodgkin's lymphoma (NHL)

  * Relapsed after or no response (no change/progressive disease) to no more than 2 adequate non-anthracycline-containing systemic chemotherapy regimens
  * At least 2 months of single-agent therapy (e.g., chlorambucil) AND/OR
  * At least 2 consecutive courses of polychemotherapy (e.g., cyclophosphamide, vincristine, and prednisone) or purine analogues
* Complete or partial remission or no change for at least 4 weeks after completion of prior therapy OR progression during one of a maximum of 2 prior therapy regimens
* CD20 positive
* At least 1 bidimensionally measurable mass
* No greater than 10,000,000/mL circulating tumor cells
* IgG levels at least 3 g/L
* No low-grade NHL transformed into intermediate- or high-grade NHL
* No symptomatic CNS lymphoma
* No bone marrow involvement only NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2.5 times ULN

Renal:

* Creatinine less than 2.5 times ULN
* BUN less than 2.5 times ULN

Cardiovascular:

* No severe cardiac disease (i.e., severe heart failure requiring symptomatic treatment)

Pulmonary:

* No severe pulmonary disease

Other:

* No severe neurologic or psychiatric disease
* No severe metabolic disease
* Not pregnant
* Fertile patients must use effective contraception
* No prior malignancy within the past 5 years except nonmelanomatous skin cancer, carcinoma in situ of the cervix, or other cancer curatively treated with surgical therapy
* HIV negative
* No uncontrolled asthma or allergy requiring steroids
* No known hypersensitivity or prior anaphylactic reaction to murine proteins or any component of study drug

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior rituximab
* No prior allogeneic or autologous peripheral blood stem cell transplantation
* Concurrent filgrastim (G-CSF) for stem cell mobilization allowed

Chemotherapy:

* See Disease Characteristics
* No prior anthracyclines or mitoxantrone
* No concurrent chemotherapy for stem cell mobilization

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 1999-05 (Actual); Primary Completion 2004-04 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Response to treatment

SECONDARY OUTCOMES:
Overall survival | from randomization
Progression Free survival | from randomization

CONTACTS AND LOCATIONS:
Overall Officials: M. H. J. Van Oers, MD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Robert Marcus, MD, Study Chair — Cambridge University Hospitals NHS Foundation Trust; Max M. Wolf, MD, Study Chair — Peter MacCallum Cancer Centre, Australia; Richard J. Klasa, MD, Study Chair — British Columbia Cancer Agency; Eva K. Kimby, MD, PhD, Study Chair — Karolinska Institutet
Locations (261):
- Australia (37):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Cancer Therapy Centre at Liverpool Hospital, Liverpool, New South Wales
  - Institute of Oncology at Prince of Wales Hospital, Randwick, New South Wales
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - St. George Hospital and Community Health Service, Sydney, New South Wales
  - Westmead Breast Centre at NSW Breast Cancer Institute, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Wesley Medical Centre, Auchenflower, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Townsville General Hospital, Townsville, Queensland
  - Royal Adelaide Hospital Cancer Centre, Adelaide, South Australia
  - Ashford Cancer Centre, Ashford, South Australia
  - Flinder Medical Centres, Bedford Park, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - St. John of God Hospital, Ballarat, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - John Fawkner Hospital, Coburg, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Garden Consulting Rooms, Mornington, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Mount Medical Centre, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital - Perth, Perth, Western Australia
- Belgium (7):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - U.Z. Gasthuisberg, Leuven
  - H. Hartziekenhuis - Roeselaere., Roeselare
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- Canada (32):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Nanaimo Cancer Clinic at Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Fraser Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre at Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital of Barrie, Barrie, Ontario
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Trillium Health Centre - Mississauga Site, Mississauga, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - St. Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital - Weston, Weston, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Hopital Notre- Dame du CHUM, Montreal, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
- Denmark (2):
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
  - Vejle Sygehus, Vejle
- National Cancer Institute of Egypt, Cairo, Egypt
- France (2):
  - Institut Bergonie, Bordeaux
  - Institut Gustave Roussy, Villejuif
- National Institute of Oncology, Budapest, Hungary
- Centro di Riferimento Oncologico - Aviano, Aviano, Italy
- Netherlands (84):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Ijselmeer Ziekenhuis - Zuiderzeeziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfont
  - St. Lucas - Andreas Ziekenhuis, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Boveny Ziekenhuis, Amsterdam
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Slotervaart Ziekenhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Albert Schweitzerziekenhuis- Zwijndrecht, Amsterdam
  - Scheperziekenhuis, Amsterdam
  - Gelre Ziekenhuizen - Lokatie Lukas, Apeldoorn
  - Ziekenhuis Lievensberg, Bergen op Zoom
  - Streekziekenhuis Gooi-Noord, Blaricum
  - Amphia Ziekenhuis - locatie Langendijk, Breda
  - Amphia Ziekenhuis - locatie Molengracht, Breda
  - Atrium Medical Centre - Brunssum, Brunssum
  - Ijsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Group - Delft, Delft
  - Gemini Ziekenhuis, Den Helder
  - Deventer Ziekenhuisen, Deventer
  - Van Weel Bethesda Ziekenhuis, Dirksland
  - NIJ Smellinghe, Drachten
  - Diaconessenhuis Eindhoven, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - St. Anna Ziekenhuis, Geldrop
  - Beatrixziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Kennemer Gasthuis - Locatie EG, Haarlem
  - Spaarne Ziekenhuis Haarlem, Haarlem
  - Ziekenhuis St Jansdal, Harderwijk
  - Tjongerschans Ziekenhuis, Heerenveen
  - Atrium Medical Centre - Heerlen, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - Streekziekenhuis Midden-Twente, Hengelo
  - Westfries Gasthuis, Hoorn
  - Zweedse Rode Kruis Ziekenhuis, La Zierikzee
  - Medisch Centrum Leeuwarden - Zuid, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Diaconessenhuis Leiden, Leiden
  - Rijnland Ziekenhuis, Leiderdorp
  - Medisch Centrum Haaglanden Antoniushove, Leidschendam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Nederlandse Hervormde Diaconessenhuisinrichting, Meppel
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen
  - Ziekenhuis Bernhoven, Oss
  - Waterlandziekenhuis, Purmerend
  - Saint Laurentius Ziekenhuis, Roermond
  - Saint Franciscus Ziekenhuis, Roosendaal
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - St. Franciscus Gasthuis, Rotterdam
  - Medisch Centrum Rynmond-Zuid - Lokatie Zuider, Rotterdam
  - Medisch Centrum Rynmond Zuid - Lokatie: Clara, Rotterdam
  - Havenziekenhiuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Maasland Hospital, Sittard
  - Albert Schweitzerziekenhuis- Sliedrecht, Sliedrecht
  - Ruwaard Van Putten Ziekenhuis, Spykenisse
  - Ziekenhuis Refaja, Stadskanaal
  - Ziekenhuis de Honte, Terneuzen
  - Hagaziekenhuis, The Hague
  - Red Cross Hospital, The Hague
  - Rivierenland Tiel, Tiel
  - St. Elisabeth Ziekenhuis, Tilburg
  - Twee Steden Ziekenhuis Vestiging Tilburg, Tilburg
  - University Medical Center Utrecht, Utrecht
  - Mesos Medisch Centrum - Overvecht, Utrecht
  - Oudenrijn Ziekenhuis, Utrecht
  - St. Joseph Veghel, Veghel
  - Maxima Medisch Centrum - locatie Eindhoven, Veldhoven
  - Holy-Ziekenhuis, Vlaardingen
  - Reinier de Graaf Group - Voorburg, Voorburg
  - St. Jans Gasthuis Weert, Weert Be
  - Hofpoort Ziekenhuis, Woerden
  - Zaans Medisch Centrum, Zaandam
  - Lorentz Ziekenhuis, Zeist
  - 'T Lange Land Ziekenhuis, Zoetermeer
  - Isala Klinieken - locatie Sophia, Zwolle
  - Isala Klinieken - locatie Weezenlanden, Zwolle
- New Zealand (3):
  - University of Auckland School of Medicine, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- Norway (3):
  - Haukeland Hospital - University of Bergen, Bergen
  - Norwegian Radium Hospital, Oslo
  - St. Olavs University Hospital, Trondheim
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon, Portugal
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Institute of Oncology - Ljubljana, Ljubljana, Slovenia
- South Africa (4):
  - Mary Potter Oncology Centre, Brooklyn Square
  - Sandton Oncology Centre, Johannesburg
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Johannesburg General Hospital, Parktown
- Sweden (8):
  - Sahlgrenska University Hospital at Gothenburg University, Gothenburg (Goteborg)
  - University Hospital of Linkoping, Linköping
  - Sunderby Hospital, Luleå
  - Lund University Hospital, Lund
  - Orebro University Hospital, Örebro
  - Karolinska University Hospital - Huddinge, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Umea Universitet, Umeå
- United Kingdom (72):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - Royal United Hospital, Bath, England
  - City Hospital - Birmingham, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Hospitals NHS Trust, Bradford, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Conquest Hospital, Canterbury, England
  - Kent and Canterbury Hospital, Canterbury, England
  - St Helier Hospital, Carshalton, England
  - Cheltenham General Hospital, Cheltenham, England
  - Countess of Chester Hospital, Chester, England
  - Essex County Hospital, Colchester, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Russells Hall Hospital, Dudley, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - Royal Free and University College Medical School, Hampstead, London, England
  - Hinchingbrooke Hospital, Huntingdon, England
  - King George Hospital, Ilford, Essex, England
  - Leeds General Infirmary at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's and St. Thomas' Hospitals NHS Foundation Trust, London, England
  - St. George's Hospital, London, England
  - St. Georges Hospital Medical School, London, England
  - Royal Marsden NHS Foundation Trust - London, London, England
  - University College Hospital, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Portsmouth Hospitals NHS Trust, Portsmouth, England
  - Whiston Hospital, Prescot Merseyside, England
  - Royal Preston Hospital, Preston, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Oldchurch Hospital, Romford, England
  - Pembury Hospital, Royal Tunbridge Wells, Kent, England
  - Salisbury District Hospital, Salisbury, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - North Staffs Royal Infirmary, Stoke-on-Trent, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Singleton Hospital, Swansea, England
  - Taunton and Somerset Hospital, Taunton Somerset, England
  - Torbay Hospital, Torquay Devon, England
  - Hillingdon Hospital, Uxbridge, England
  - Sandwell General Hospital, West Bromwich, England
  - Royal Hampshire County Hospital, Winchester, England
  - New Cross Hospital, Wolverhampton, England
  - Belfast City Hospital Trust, Belfast, Northern Ireland
  - Western General Hospital, Edinburgh, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - University Hospital of Wales, Cardiff, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - Glan Clywd District General Hospital, Rhyl, Denbighshire, Wales
  - Saint Richards Hospital, Chichester
  - Hull Royal Infirmary, Hull
  - Kettering General Hosptial, Kettering, Northants
  - Staffordshire General Hospital, Stafford
  - Great Western Hospital, Swindon

REFERENCES:
- [Background] Deconinck E, Miadi-Fargier H, Pen CL, Brice P. Cost effectiveness of rituximab maintenance therapy in follicular lymphoma: long-term economic evaluation. Pharmacoeconomics. 2010;28(1):35-46. doi: 10.2165/11314070-000000000-00000. PMID 20014875
- [Background] Pompen M, Huijgens PC, et al.: Cost-effectiveness of rituximab for maintenance in patients with follicular non-Hodgkin's lymphoma in the Dutch setting. [Abstract] Blood 112 (11): A-2364, 2008.
- [Background] Van Oers MH, Hagenbeek A, Van Glabbeke M, Teodorovic I. Chimeric anti-CD20 monoclonal antibody (Mabthera) in remission induction and maintenance treatment of relapsed follicular non-Hodgkin's lymphoma: a phase III randomized clinical trial--Intergroup Collaborative Study. Ann Hematol. 2002 Oct;81(10):553-7. doi: 10.1007/s00277-002-0548-2. Epub 2002 Oct 17. No abstract available. PMID 12424535
- [Result] van Oers MH, Tonnissen E, Van Glabbeke M, Giurgea L, Jansen JH, Klasa R, Marcus RE, Wolf M, Kimby E, Vranovsky A, Holte H, Hagenbeek A, van der Reijden BA. BCL-2/IgH polymerase chain reaction status at the end of induction treatment is not predictive for progression-free survival in relapsed/resistant follicular lymphoma: results of a prospective randomized EORTC 20981 phase III intergroup study. J Clin Oncol. 2010 May 1;28(13):2246-52. doi: 10.1200/JCO.2009.25.0852. Epub 2010 Apr 5. PMID 20368567
- [Result] van Oers MH, Van Glabbeke M, Giurgea L, Klasa R, Marcus RE, Wolf M, Kimby E, van t Veer M, Vranovsky A, Holte H, Hagenbeek A. Rituximab maintenance treatment of relapsed/resistant follicular non-Hodgkin's lymphoma: long-term outcome of the EORTC 20981 phase III randomized intergroup study. J Clin Oncol. 2010 Jun 10;28(17):2853-8. doi: 10.1200/JCO.2009.26.5827. Epub 2010 May 3. PMID 20439641
- [Result] van Oers MH, Klasa R, Marcus RE, Wolf M, Kimby E, Gascoyne RD, Jack A, Van't Veer M, Vranovsky A, Holte H, van Glabbeke M, Teodorovic I, Rozewicz C, Hagenbeek A. Rituximab maintenance improves clinical outcome of relapsed/resistant follicular non-Hodgkin lymphoma in patients both with and without rituximab during induction: results of a prospective randomized phase 3 intergroup trial. Blood. 2006 Nov 15;108(10):3295-301. doi: 10.1182/blood-2006-05-021113. Epub 2006 Jul 27. PMID 16873669
- [Derived] Mattiola I, Mantovani A, Locati M. The tetraspan MS4A family in homeostasis, immunity, and disease. Trends Immunol. 2021 Sep;42(9):764-781. doi: 10.1016/j.it.2021.07.002. Epub 2021 Aug 9. PMID 34384709